CLINICAL TRIAL: NCT06392165
Title: Evaluation of Adhesion Properties in Wound Care Devices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DNR-2024-00715-02
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Adhesion Properties of Wound Care Devices

STUDY DESIGN:
Intervention Model Description: intra-individual test with up 12 test samples per study run; this treatment is announced here as single group study.
Masking Description: all participants will receive the same up to 12 test samples, which are randomized intra-individual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-adhesive wound care devices (Other): test devices with adhesive material to be attached to skin
  Interventions: Other: self-adhesive device

INTERVENTIONS:
Other: self-adhesive device — Test device which is self-adhesive

SUMMARY:
Molnlycke manufactures and markets self-adhesive wound care devices intended to protect various types of wounds during treatment. This study aims to measure and evaluate the adhesion properties of self-adhesive wound care devices. To measure the adhesion properties test strips will be applied to the participant's skin for a predetermined time and will be removed while measuring the adhesion properties afterwards. This method has been chosen since there is no in vitro method available that can simulate adhesion to human skin

ELIGIBILITY:
Inclusion Criteria:

* Confirmed eligibility and signed consent form.

Exclusion Criteria:

* Known plaster allergy or other known contact hypersensitivity
* Pregnant or breastfeeding individual.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-24 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Peel Off Force | up to 48 hours
  Internal machine shall measure the peel force expressed in Newton.

SECONDARY OUTCOMES:
Humidity | up to 48 hours
  Humidity shall be evaluated using tactile and visual assessment
Redness | up to 48 hours
  Visual assessment of redness of the skin
Pain assessment | up to 48 hours
  Visual analog scale (VAS) assessment of pain after removal. The scale is 100mm long whether 0mm means no pain and 100mm means the maximum pain a participant could imagine.

OTHER OUTCOMES:
Adhesive residuals | up to 48 hours
  Adhesive residuals on the skin
Loosening | up to 48 hours
  Assessment if the device is still in place or has been fallen of.
Comments | up to 48 hours
  Further comments (not related to the other outcomes) by the participant or the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Mölnlycke Health Care AB, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No